CLINICAL TRIAL: NCT06493799
Title: A Multicenter, Randomized, Open-label, Active-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Intravenous Drop of 'LAENNEC INJ. (Human Placenta Hydrolysate) Compared With Subcutaneous Injection in Patients With Chronic Liver Disease
Brief Title: In Patients With Chronic Liver Diseases(Alcoholic Liver Disease and Non-Alcoholic Fatty Liver Disease), LAENNEC(Human Placenta Hydrolysate) is to Evaluate the Efficacy and Safety of Intravenous Drop
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Wellbeing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAEN-IV3
Record Dates: First submitted 2024-06-30; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAENNEC 10 ml(Intravenous Injection) (Experimental): Dosing twice a week for 6 weeks
  Interventions: Drug: LAENNEC (Human Placenta Hydrolysate) IV
- LAENNEC 4 ml(Subcutaneous Injection) (Active Comparator): Dosing twice a week for 6 weeks
  Interventions: Drug: LAENNEC (Human Placenta Hydrolysate) SC

INTERVENTIONS:
Drug: LAENNEC (Human Placenta Hydrolysate) IV — Intravenous Injection
  Arms: LAENNEC 10 ml(Intravenous Injection)
Drug: LAENNEC (Human Placenta Hydrolysate) SC — Subcutaneous Injection
  Arms: LAENNEC 4 ml(Subcutaneous Injection)

SUMMARY:
Control group : LAENNEC subcutaneous injection (4 ml)

Experimental group : LAENNEC intravenous injection (10 ml)

DETAILED DESCRIPTION:
This is a multi- center, randomized, open-label, Active-controlled phase 3 trial in participants aged 18 to 70 years with chronic liver disease. It is designed to assess the safety, tolerability and efficacy of both 4 ml SC and 10ml IV LAENNEC when administered twice of week for 6 weeks. A total of 226 participants will be randomised to received 4ml SC or 10ml IV of LAENNEC a 1:1 ratio. And in 4 ml SC and 10 ml IV, the ratio of ALD and NAFLD is 1:3. The investigational product will be administered SC or IV twice of week for a duration of 6 weeks. Participants will return to the clinic for follow-up safety and efficacy assessments on weeks 2, 4, 6.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for participation in the trial if all of the following inclusion criteria are met:

1. At the time of screening, 19 or 70 years
2. Those who have been diagnosed with alcoholic or non-alcoholic fatty liver disease
3. Those who have increased ALT level (Increased ALT level : 60 IU/L ≤ ALT ≤ 200 IU/L)
4. A person who can complete the signature agreement and comply with clinical trial requirements.

Exclusion Criteria:

A participant will not be eligible for trial participation if any of the following exclusion criteria are met:

1. If you have the following disease

   * Liver cancer or other malignant tumor within 5 years at screening point
   * Esophageal varix bleeding, hepatic coma, ascites etc. related disease or Child-Pugh Score Class B,C patient within 1 year at screening point
   * Organs or bone marrow transplant experience
   * Billiary atresia, Genetic metabolic liver disease, Fulminant Hepatic failure, toxicity or Clinically diagnosed hepatitis, bleeding or Platelet disease patient
   * Autoimmune hepatitis, Primary biliary cirrhosis, Sclerosing cholangitis, IgG4- associated cholangitis patient
   * Bariatric Surgery within 24 weeks at screening point
   * Uncontrolled diabetes mellitus (HBA1c > 9.0%)
   * Uncontrolled serious Cardiopulmonary disease
   * Liver cancer or other malignant tumor within 5 years at screening point
   * Those who have alcohol abuse within 5 years at screening point
   * Hepatitis B, C virus (However, those who have been identified as HBV DNA undetectable or SVR after antiviral administration can participate)
   * Systemic infection (including tuberculosis)
2. If you are taking the following drug (Hepatotonics)

   * However, it is possible to register after having a drug holiday

     * Biphenyl dimethyl dicarboxylate (BDD), Silymarin(Milk thistle) : 14 days
     * Ursodeoxycholic acid (UDCA) : 30 days
     * Other Hepatotonics : 5 times half-life
3. If you are taking the following drug or need to take drugs during the clinical trial period

   * Antituberculous drug(Isoniazid, Rifampin etc.), antifungal agent and antibiotic
   * Acetaminophen, NSAIDs(Excluding low-dose aspirin for preventive purposes)
   * Lipid lowering agent(Niacin etc.) and Oral hypoglycemic agent(acarbose etc.) (Registered when administered during the clinical trial period with a certain dose without a change in dose currently being taken)
   * Antiseric agent (ARB, Beta-blocker, CCB etc.) (Registered when administered during the clinical trial period with a certain dose without a change in dose currently being taken)
   * Vitamin E (Purpose of treatment of more than 800 IU/day)
   * Astrogens
   * Systemic corticosteroids, Immunomodulator
4. If you take more alcohol than the recommended amount (Man 40 g/day, Woman 20 g/day)
5. Drug allergic symptoms (oscillation, heat, itching)
6. Those who have received other clinical drugs within 4 weeks before selecting a test subject
7. Those who cannot inject intravenous infusions (5% Dextrose Inj.)
8. A person who does not perform appropriate contraception as a pregnant woman, a nursing or a woman of childbearing age (effective contraception method: Barrier methods using infertility surgery, uterine device, condom, killer)
9. Those who judged that other testors were inappropriate as clinical trials

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ALT level relative to baseline at 6 weeks | week 6
  In order to compare the test groups and control groups, check the ALT change after 6 weeks compared to the baseline.
  For the 6 week ALT change amount, a civic analysis (ANCOVA) is performed with the ALT level of the base line and the tamed dynasty (alcohol liver disease/non -alcohol liver liver disease) in a covenant.
  In addition, depending on the normal distribution of the data, the Paired t-test or Wilcoxon's rank test is performed to confirm the difference in the average change in the military.

SECONDARY OUTCOMES:
Change in ALT level relative to baseline at 2, 4 weeks | week 2, 4
  In order to compare the test groups and control groups, check the ALT change after 2,4 weeks compared to the baseline.
  For the 2,4 weeks ALT change amount, a civic analysis (ANCOVA) is performed with the ALT level of the base line and the tamed dynasty (alcohol liver disease/non -alcohol liver liver disease) in a covenant.
  In addition, depending on the normal distribution of the data, the Paired t-test or Wilcoxon's rank test is performed to confirm the difference in the average change in the military.
Change in AST, Total Bilirubin and r-GT level relative to baseline at 2, 4, 6 weeks | week 2, 4, 6
  In order to compare the test groups and control groups, check the AST, Total Bilirubin and r-GT change after 2,4,6 weeks compared to the baseline.
  For the 2, 4, 6 weeks AST, Total Bilirubin and r-GT change amount, a civic analysis (ANCOVA) is performed with the ALT level of the base line and the tamed dynasty (alcohol liver disease/non -alcohol liver liver disease) in a covenant.
  In addition, depending on the normal distribution of the data, the Paired t-test or Wilcoxon's rank test is performed to confirm the difference in the average change in the military.
The rate of ALT normalization at 2, 4, 6 weeks | week 2, 4, 6
  Check the difference by conducting Chi-Square Test or Fisher's Exact Test for the number and ratio of the ALT normal level at 2, 4, 6 weeks.
The rate of AST normalization at 2, 4, 6 weeks | week 2, 4, 6
  Check the difference by conducting Chi-Square Test or Fisher's Exact Test for the number and ratio of the AST normal level at 2, 4, 6 weeks.
ALT normalization time | during 6 week
  It presents the time to normalize the ALT of the test group and the control group, and checks the difference between the test group and the control group using the log order test.
The Rate of participants with ≤ 20% decrease of ALT relative to baseline at 2, 4 weeks | week 2, 4, 6
  Check the difference by conducting Chi-Square Test or Fisher's Exact Test for the number and ratio of the ≤ 20% decrease of ALT relative to baseline at 2, 4, 6 weeks.
Change in FSS score relative to baseline at 6 weeks | week 6
  In order to compare the test groups and control groups, check the FSS change after 6 week compared to the baseline.
  For the 6 week FSS change amount, a civic analysis (ANCOVA) is performed with the ALT level of the base line and the tamed dynasty (alcohol liver disease/non -alcohol liver liver disease) in a covenant.
  In addition, depending on the normal distribution of the data, the Paired t-test or Wilcoxon's rank test is performed to confirm the difference in the average change in the military.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Up Kim, Ph.D., Study Director — 50-1, Yonsei-ro, Seodaemun-gu, Seoul, Republic of Korea; Eileen Laurel Yoon, Ph.D., Study Director — 222-1, Wangsimni-ro, Seongdong-gu, Seoul, Republic of Korea; Sang Gyune Kim, Ph.D., Study Director — 170, Jomaru-ro, Wonmi-gu, Bucheon-si, Gyeonggi-do, Republic of Korea; Yuri Cho, Ph.D., Study Director — 323, Ilsan-ro, Ilsandong-gu, Goyang-si, Gyeonggi-do, Republic of Korea; Jung Hwan Yu, Ph.D., Study Director — 27, Inhang-ro, Jung-gu, Incheon, Republic of Korea; Won Sohn, Ph.D., Study Director — 29, Saemunan-ro, Jongno-gu, Seoul, Republic of Korea; Soo Young Park, Ph.D., Study Director — 807, Hoguk-ro, Buk-gu, Daegu, Republic of Korea; Byoung Kuk Jang, Ph.D., Study Director — 1035, Dalgubeol-daero, Dalseo-gu, Daegu, Republic of Korea; Soung Won Jeong, Ph.D., Study Director — 59, Daesagwan-ro, Yongsan-gu, Seoul, Republic of Korea; Young Youn Cho, Ph.D., Study Director — 102, Heukseok-ro, Dongjak-gu, Seoul, Republic of Korea; Eun Ju Cho, Ph.D., Study Director — 101, Daehak-ro, Jongno-gu, Seoul, Republic of Korea; Jung Gil Park, Ph.D., Study Director — 70, Hyeonchung-ro, Nam-gu, Daegu, Republic of Korea; Jung Hyun Kwon, Ph.D., Study Director — 56, Dongsu-ro, Bupyeong-gu, Incheon, Republic of Korea; Young Kul Jung, Ph.D., Study Director — 123, Jeokgeum-ro, Danwon-gu, Ansan-si, Gyeonggi-do, Republic of Korea; Ja Kyung Kim, Ph.D., Study Director — 363, Dongbaekjukjeon-daero, Giheung-gu, Yongin-si, Gyeonggi-do, Republic of Korea; Hyun Woong Lee, Ph.D., Study Director — 211, Eonju-ro, Gangnam-gu, Seoul, Republic of Korea; Won Hyeok Choe, Ph.D., Study Director — 120-1, Neungdong-ro, Gwangjin-gu, Seoul, Republic of Korea; Chun Kyon Lee, Ph.D., Study Director — 100, Ilsan-ro, Ilsandong-gu, Goyang-si, Gyeonggi-do, Republic of Korea